CLINICAL TRIAL: NCT05633290
Title: CharacterisatiON of carDiac funCTion in Intensive Care Unit Survivors of Sepsis (CONDUCT-ICU): A Pilot Study
Brief Title: CharacterisatiON of carDiac funCTion in Intensive Care Unit Survivors of Sepsis.
Acronym: CONDUCT-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: NHS Ayrshire and Arran (Other); Golden Jubilee National Hospital (Other Government); University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN22CA029
Record Dates: First submitted 2022-03-14; First posted 2022-12-01 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Myocarditis; Sepsis; Septic Shock
MeSH Terms: conditions — Heart Failure; Myocarditis; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Survivors of Sepsis: ICU survivors of sepsis who would routinely attend ICU follow-up.
  Interventions: Diagnostic Test: CMR; Diagnostic Test: hs-troponin; Diagnostic Test: NT-pro BNP; Diagnostic Test: CRP; Diagnostic Test: IL1-B; Diagnostic Test: IL-6; Diagnostic Test: IL-10; Diagnostic Test: TNF-alpha

INTERVENTIONS:
Diagnostic Test: CMR — CMR Imaging 6-10 weeks post hospital discharge.
Diagnostic Test: hs-troponin — Biomarker of myocardial injury
Diagnostic Test: NT-pro BNP — Biomarker for heart failure
Diagnostic Test: CRP — Acute phase inflammatory marker
Diagnostic Test: IL1-B — Inflammatory biomarker
Diagnostic Test: IL-6 — Inflammatory Biomarker
Diagnostic Test: IL-10 — Inflammatory Biomarker
Diagnostic Test: TNF-alpha — Inflammatory Biomarker

SUMMARY:
Cardiac dysfunction is common following hospital admission with sepsis and one of the most frequent causes for readmissions to hospital, however underlying mechanisms by which this might occur are unclear. The CONDUCT-ICU investigators will conduct a pilot, cohort study, characterizing cardiac function in ICU survivors of sepsis using a combination of CMR imaging, biomarkers and patient reported outcome measures to investigate mechanisms of cardiac dysfunction following sepsis. Comparisons will be made to that of the general population.

DETAILED DESCRIPTION:
Sepsis is one of the most common reasons for admission to ICU in the UK and it is well established that adverse cardiovascular events are common following sepsis. In fact, the risk of adverse cardiovascular events such as MI, Heart Failure and Stroke is in excess of 60% greater compared to those who have not had sepsis. Similarly, heart failure is one of the most common causes of readmission to hospital following an episode of sepsis. The underlying mechanisms for this phenomenon are unclear and CONDUCT-ICU investigators intend on answering this question.

Investigators will collect cardiac and inflammatory biomarkers from participants at the point of discharge from ICU. Following discharge from hospital, cardiac magnetic resonance (CMR) scans of the heart will be undertaken in participants 6-10 weeks post-discharge from hospital to examine for evidence of inflammation in the heart. Further blood samples will also be collected to look for evidence of inflammation and heart muscle injury at this point in addition to patient reported outcomes measures using validated questionnaires.

Participants will be identified with their direct clinical team in ICU and are nearing or at the point of discharge from ICU. If eligible for the study, they will be approached by researchers and provided them with an information sheet and written consent form. Participants will be given up to 24hrs to decide if they wish to take part in research and if so, they will sign the consent form. Participants are free to withdraw from the study at any time, without any reason given, and this would not affect the standard of care they receive.

This is an observational cohort study. If willing to take part, participants will receive the normal follow-up that would be undertaken following discharge from ICU. In addition, researchers will collect a sample of blood from participants at the time of discharge from ICU and again at 6 -10 weeks post discharge. A Cardiac Magnetic Resonance (CMR) scan will be undertaken 6-10 weeks follow up.

Researchers will assess the patient's day-to-day function and quality of life by asking them to complete validated questionnaires. These questionnaires should take five to ten minutes to complete and help will be available if required. Participants will complete these questionnaires at the follow-up visit 6-10 weeks following discharge from hospital with the help of the researchers conducting the study

The first blood sample will be collected following discharge from ICU whilst the patient is still in hospital. Further blood samples will be collected 6-10 weeks following discharge from hospital. Blood samples for patients undergoing CMR will be taken when they attend for scan. Blood sampling for patients who do not undergo CMR imaging will attend for a separate follow-up visit for collection of samples.

Patients are normally invited to attend ICU follow-up via the InS:PIRE service at approximately 6-10 weeks post-discharge. Where possible researchers will combine blood sample analysis with routine follow-up visits in clinic to which participants would normally be invited. If they are not able to attend follow-up and are not attending for CMR scan, then researchers will invite them to the research facility within the local sites for collection of samples.

Samples will be stored in NHS Biorepository and analyzed within the British Heart Foundation Laboratory at the University of Glasgow.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Age > 18 years.
3. ICU admission with sepsis (According to The Third International Consensus Definitions for Sepsis and Septic Shock [Sepsis-3])17
4. Ability to comply with study procedures

Exclusion Criteria:

1. Inability to give informed consent
2. Pregnancy.
3. Ongoing participation in any investigational research that may undermine the scientific basis of the study.
4. Contraindications to magnetic resonance imaging:

   i. Cardiac pacemaker, artificial heart valve, neurostimulator, cochlear implant ii. Aneurysm clips iii. Metal injuries to the eye iv. Loose metal in any part of the body v. Severe claustrophobia
5. Known Coronary Artery Disease
6. Previous Myocardial Infarction
7. Chronic Heart Failure prior to ICU admission
8. Patient receiving immune modulating drug or biologic therapy either long term or during acute admission
9. Patient considered by the clinical team to be very unlikely to survive to hospital discharge
10. Hospital Admission because of Covid-19
11. Patients undergoing treatment for malignancy with systemic anti-cancer therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU Survivors of Sepsis
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction | 6-10 weeks post hospital discharge
  LVEF is a validated marker of cardiovascular function. It can be used in diagnosis of heart failure and can assist in grading severity.

SECONDARY OUTCOMES:
hs-Troponin (ng/L) | 6-10 weeks post-hospital discharge
  Marker of myocardial injury commonly used in clinical practice
NT-proBNP (pg/ML) | 6-10 weeks post-hospital discharge
  Biomarker of myocardial dysfunction used in patients with heart failure and associated conditions.
CRP (mg/L) | 6-10 weeks post discharge
  Acute phase biomarker of inflammation.
IL-10 (pg/ml) | 6-10 weeks post discharge
  Inflammatory cytokine thought to inhibit innate immune response.
IL-1B (pg/ml) | 6-10 weeks post discharge
  Acute phase inflammatory cytokine and pyrogen.
TNF-alpha (pg/ml) | 6-10 weeks post discharge
  Inflammatory cytokine implicated in acute inflammation and targeted for management of inflammatory and autoimmune disease
IL-6 (pg/ml) | 6-10 weeks post discharge
  Inflammatory biomarker associated with adverse cardiovascular outcomes and adverse mortality in critically ill patients
Brief Pain Inventory Score | 6-10 weeks post discharge
  Validated Assessment of Pain. Scores of 0 indicate no pain and scores of 10 indicate the 'worst pain you can imagine'.
ID Pain Score | 6-10 weeks post discharge
  Validated assessment tool for differentiation of neuropathic pain. Patients describe character of pain using 'yes' or 'no' questions.
EuroQol 5-Dimension (5D) Score | 6-10 weeks post discharge
  Validated measure of quality of life. Part of core outcome measures in critical illness survivors. Scores 5 domains (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety /Depression) on likert scale as follows: 1) No problems, 2) Slight Problems, 3) Moderate Problems, 4) Severe Problems, 5) Unable
Hospital Anxiety and Depression Score | 6-10 weeks post discharge
  Validated measure of anxiety and depression. Previously used in survivors of critical illness. Total score: 0-7 = Normal, 8-10 Borderline abnormal (borderline case), 11-21 Abnormal (case)
Dukes Activity Status Index | 6-10 weeks post discharge
  Validated tool for assessing functional capacity. Scores 0 - 58.2, with higher scores indicating better functional capacity.
Vitality Domain of Short Form 36 - Score | 6-10 weeks post discharge
  Validated tool for vitality and used in survivors of critical illness. Likert Scale Assessing vitality. Answers range from 1)All of the time, most of the time, a good bit of the time, some of the time, a little bit of the time, none of the time.
MRC Breathlessness Scale | 6-10 weeks post discharge
  Widely used grading system for breathlessness in survivors of critical illness. Graded 0-4.4 indicates more severe breathlessness.
Myocardial Native T1 and T2 Mapping | 6-10 weeks post discharge
  CMR markers of subtle inflammation and fibrosis commonly examined during CMR imaging.
Successful follow-up rate of participants invited to attend CMR scans. i.e. Feasibility of CMR imaging | 6-10 weeks post discharge
  To evaluate feasibility of undertaking CMR in complex post-ICU cohort of patients. To the investigators' best knowledge, this cohort has never been investigated before in this way and it is unclear to what extent participants will be able to attend follow up. We will evaluate the attendance rate at CMR follow-up measured against participants invited to take part in the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Glasgow Royal Infirmary, Glasgow
  - University Hospital Crosshouse, Kilmarnock

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrity K, Docherty C, Mangion K, Woodward R, Shaw M, Roditi G, Shelley B, Quasim T, McCall P, McPeake J. Characterizing Cardiac Function in ICU Survivors of Sepsis: A Pilot Study Protocol. CHEST Crit Care. 2024 Mar;2(1):100050. doi: 10.1016/j.chstcc.2024.100050. PMID 38524255